CLINICAL TRIAL: NCT02220335
Title: Pulmonary Arterial Denervation in Patients With Pulmonary Hypertension Associated With the Left Heart Failure: a Randomised Controlled Trial
Brief Title: Pulmonary Arterial Denervation in Patients With Pulmonary Hypertension Associated With the Left Heart Failure
Acronym: PADN-5
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Shaoliang Chen, Vice President, Nanjing First Hospital, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20140618
Record Dates: First submitted 2014-08-08; First posted 2014-08-19 (Estimated); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Pulmonary Hypertension
Keywords: pulmonary hypertension; pulmonary arterial denervation; left heart failure; 6-min walk distance
MeSH Terms: conditions — Hypertension, Pulmonary; Heart Failure | interventions — Diuretics; Angiotensin-Converting Enzyme Inhibitors; Digoxin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pulmonary Arterial Denervation (PADN) (Experimental): Contrast pulmonary artery （PA) angiography was performed to localize the pulmonary artery bifurcation level and calculate the PA diameter.Once the anatomy was deemed acceptable, the radiofrequency ablation catheter was introduced into ostium of the left PA, ostium of the right PA , and the distal bifurcation area of the main PA.This was then maneuvered within the PA to allow energy delivery in a circumferential manner to ensure that the electrodes were tightly in contact with the endovascular surface. About four to eight ablations at 10 W for 60 seconds each were performed in ostium of the left PA, ostium of the right PA , and the distal bifurcation area of the main PA.
  Interventions: Procedure: Pulmonary arterial denervation; Drug: Standard treatment
- Standard treatment (Active Comparator): Patients in the standard treatment group will take their baseline anti-heart failure medications at the original doses, without any changes except when medically required.The anti-heart failure drugs treatment is consistent in both arms.
  Interventions: Drug: Standard treatment

INTERVENTIONS:
Procedure: Pulmonary arterial denervation — Contrast pulmonary artery （PA) angiography was performed to localize the pulmonary artery bifurcation level and calculate the PA diameter.Once the anatomy was deemed acceptable, the radiofrequency ablation catheter was introduced into the distal bifurcation area of the main PA.This was then maneuvered within the PA to allow energy delivery to ensure that the electrodes were tightly in contact with the endovascular surface. About two to three ablations at 1-15 W for 240 seconds each point were performed in the distal bifurcation area of the main PA.
  Other Names: PADN
  Arms: Pulmonary Arterial Denervation (PADN)
Drug: Standard treatment — Patients in the standard treatment group will take their baseline anti-heart failure medications at the original doses, without any changes except when medically required.The anti-heart failure drugs treatment is consistent in both arms.Patients in the standard treatment group will take one or combination of the following target drugs: endothelin receptor antagonist, 5'-PDE and prostacyclin. On the other hand, patients in the PADN group do not take any of the target drugs mentioned above.
  Other Names: Diuretics; Nitrate esters; β-blockers; ACE inhibitors or receptor blockers aldosterone antagonists; Digoxin

SUMMARY:
A number of 100 patients with pulmonary hypertension associated with the left Heart failure scheduled for elective pulmonary arterial denervation (PADN) are randomized 1:1 to either PADN or control group.

DETAILED DESCRIPTION:
Heart failure patients must have completed the right heart catheterization. All the patients accepted the optimal medical therapies,including diuretics, Nitrate esters, β-blockers, ACE inhibitors or receptor blocker aldosterone antagonists and/or digoxin).The patients of pulmonary hypertension are defined into two groups: "passive" pulmonary hypertension(mPAP≥25 mmHg, PCWP>15 mmHg and pulmonary vascular resistance<3 woods unit) increase due to backward transmission of increased left ventricular filling pressure, "reactive" pulmonary hypertension (mPAP≥25 mmHg, PCWP>15 mmHg and pulmonary vascular resistance >3 woods unit) increase in resistance due to either pulmonary vasoconstriction or structural changes in the pulmonary vasculature.

All the "reactive" pulmonary hypertension patients are eligible for the randomized study in PADN group or control group according to the computer generated random table.

ELIGIBILITY:
Inclusion Criteria:

* Age>18yr
* "Reactive"Pulmonary Hypertension in Left Heart Failure: mPAP≥25 mmHg, PCWP>15 mmHg and pulmonary vascular resistance (PVR) [The PVR =(mPAP-PCWP)/ carbon monoxide]>3.0 woods unit
* Voluntary acceptance of all follow-up assessment of program requirements.

Exclusion Criteria:

* WHO group I, III, IV, V pulmonary artery hypertension
* Severe Renal dysfunction (Ccr<30 ml/min)
* Blood platelet count<100,000/L
* Expected life span<12-month
* In pregnancy
* Systematical inflammation
* Malignant cancer(s)
* Tricuspid valve stenosis, Supra-pulmonary valve stenosis
* Allergic to studied drugs or metal materials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2014-08-08 (Actual); Primary Completion 2018-06-16 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
6-min-walk distance increase | 6 months
  The primary effectiveness endpoint is change in 6-min-walk distance (6-MWD) from baseline to 6 months post-randomization.

SECONDARY OUTCOMES:
Pulmonary vascular resistance | 6 months
  Measure pulmonary vascular resistance using 2D doppler echocardiogram w/definity. Correlation coefficients between the technique above the the gold standard right heart catheterization measures of pulmonary vascular resistance.

OTHER OUTCOMES:
Accuracy of pulmonary embolism | 6 months
  The safety endpoint is the accuracy of pulmonary embolism (PE). Suspected PE with one of the following:
  1. new intra-luminal filling defect on CT scan, MRI scan, or pulmonary angiogram;
  2. new perfusion defect of at least 75% on V/Q lung scan;
  3. inconclusive spiral CT, pulmonary angiography or lung scan with demonstration of deep vein thrombosis in the lower extremities by venography
  Fatal PE is:
  1. PE based on objective diagnostic testing or autopsy or
  2. death not attributed to a documented cause and for which deep vein thrombosis/PE cannot be ruled out.

CONTACTS AND LOCATIONS:
Overall Officials: Shaoliang Chen, MD, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang H, Kan J, Zhang J, Xie D, Li X, Zhou W, Dong J, Gu H, Han Y, Chen SL. 3-Year Outcome in Patients With Combined Precapillary and Postcapillary Pulmonary Hypertension: Results From PADN-5 Trial. JACC Heart Fail. 2023 Aug;11(8 Pt 2):1135-1146. doi: 10.1016/j.jchf.2023.05.016. Epub 2023 Jun 21. PMID 37354146
- [Derived] Zhang H, Zhang J, Chen M, Xie DJ, Kan J, Yu W, Li XB, Xu T, Gu Y, Dong J, Gu H, Han Y, Chen SL. Pulmonary Artery Denervation Significantly Increases 6-Min Walk Distance for Patients With Combined Pre- and Post-Capillary Pulmonary Hypertension Associated With Left Heart Failure: The PADN-5 Study. JACC Cardiovasc Interv. 2019 Feb 11;12(3):274-284. doi: 10.1016/j.jcin.2018.09.021. Epub 2018 Oct 23. PMID 30732732